CLINICAL TRIAL: NCT00477867
Title: Assessing Economic Outcomes in Women With Stage III Ovarian Cancer Treated With Intravenous Paclitaxel and Cisplatin v. Intravenous Paclitaxel, Intraperitoneal Cisplatin and Intraperitoneal Paclitaxel on GOG #172: A Feasibility Study of Assessing Costs and Medical Resource Use
Brief Title: Economic Outcomes in Patients With Stage III Ovarian Cancer Receiving Paclitaxel and Cisplatin on Clinical Trial GOG-172
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was never activated
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Health Services Research
Other Study IDs: CDR0000078639; GOG-9905
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2007-10

CONDITIONS: Ovarian Cancer
Keywords: stage III ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

INTERVENTIONS:
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Gathering information about patients with ovarian cancer over time may help doctors learn more about a patient's use of medical services and the cost of these services.

PURPOSE: This clinical trial is collecting information about the patient's health and use of medical resources over time in patients with stage III ovarian cancer receiving paclitaxel and cisplatin on clinical trial GOG-172.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of collecting data on medical resource utilization and costs incurred in the care of patients with stage III ovarian cancer treated with intravenous (IV) paclitaxel and cisplatin vs IV paclitaxel, intraperitoneal (IP) paclitaxel, and IP cisplatin on a randomized, controlled clinical trial.
* Determine the feasibility of collecting data on resource utilization incurred outside GOG institutions through the use of patient diaries.
* Assess the work load required to collect this data, in terms of mean number of hours required to complete medical resource utilization forms.

OUTLINE: Data on medical resource units consumed (including length of hospital stay, length of time using operating room, units of drugs and blood products administered, number of diagnostic tests received, and number of physician visits needed) are collected on all patients.

Quality of life is assessed prior to randomization on clinical trial GOG-172, prior to the fourth course of chemotherapy, after the sixth course of chemotherapy, and at 3 months and 6 months after the sixth course of chemotherapy. Patients complete diaries throughout treatment with chemotherapy and for 12 months after treatment.

Data collected are used for analysis of economic impact, quality of life, neurotoxicity, and sociologic characteristics associated with these treatment regimens.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage III ovarian cancer
* Concurrent enrollment on clinical trial GOG-172 required

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* GOG 0-3

Life expectancy:

* Not specified

Other:

* Able to communicate in English or Spanish

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Feasibility of collecting data on medical resource utilization and costs incurred in the care of patients with stage III ovarian cancer
Feasibility of collecting data on resource utilization incurred outside GOG institutions
Work load required to collect this data, in terms of mean number of hours required to complete medical resource utilization forms

CONTACTS AND LOCATIONS:
Overall Officials: Martee L. Hensley, MD, Study Chair — Memorial Sloan Kettering Cancer Center